CLINICAL TRIAL: NCT07123441
Title: A Study on the Efficacy and Safety of Irinotecan Liposome (II), 5-FU/LV in Combination With Bevacizumab for the Treatment of Advanced Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanjun Cai (Other)
Responsible Party: Sponsor-Investigator, Sanjun Cai, professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDCRC108-CSJ
Record Dates: First submitted 2025-08-01; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer， irinotecan liposome (II)，5-FU/LV
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): Bevacizumab: 5 mg/kg, intravenous infusion, Day 1; Irinotecan liposome (II): 60 mg/m² (based on free base), intravenous infusion for at least 90 minutes, Day 1 ; 5-FU: 400 mg/m², intravenous bolus injection, Day 1; followed by 1200 mg/(m²·day) × 2 days of continuous intravenous infusion (total dose 2400 mg/m², infused over 46-48 hours); LV: 400 mg/m², intravenous infusion over 2 hours, Day 1; Q2w, continued until an event meeting the treatment discontinuation criteria occurs or the subject withdraws from the study.
  Interventions: Drug: Bevacizumab,Irinotecan liposome (II),5-FU/LV

INTERVENTIONS:
Drug: Bevacizumab,Irinotecan liposome (II),5-FU/LV — Bevacizumab: 5 mg/kg, intravenous infusion, Day 1; Irinotecan liposome (II): 60 mg/m² (based on free base), intravenous infusion for at least 90 minutes, Day 1; 5-FU: 400 mg/m², intravenous bolus injection, Day 1; followed by 1200 mg/(m²·day) × 2 days of continuous intravenous infusion (total dose 2400 mg/m², infused over 46-48 hours); LV: 400 mg/m², intravenous infusion over 2 hours, Day 1; Q2w, continued until an event meeting the treatment discontinuation criteria occurs or the subject withdraws from the study.

SUMMARY:
This is a single-arm, open-label clinical trial designed to evaluate the efficacy and safety of irinotecan liposome (II), 5-FU/LV in combination with bevacizumab for the treatment of advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, no gender restrictions;
2. Patients with pathologically confirmed, unresectable advanced colorectal cancer;
3. According to the RECIST 1.1 criteria, patients must have at least one measurable target lesion;
4. ECOG performance status: 0-1 points;
5. Expected survival period ≥3 months;
6. Good major organ function, i.e., relevant laboratory parameters within 14 days prior to randomization meet the following requirements:

(1) Complete blood count (no blood transfusion or use of leukocyte or platelet-enhancing agents within 14 days prior to screening): hemoglobin > 90 g/L; neutrophil count > 1.5 × 10⁹/L; platelet count > 100 × 10⁹/L;(2) Biochemical tests: total bilirubin ≤ 1.5×ULN (upper limit of normal); alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2×ULN; if liver metastasis is present, ALT and AST ≤ 5×ULN; endogenous creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula); (3) Cardiac Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥ 50%.

7. Any damage caused by other treatments has recovered; 8. The subject voluntarily participates in this study, has signed an informed consent form, has good compliance, and cooperates with follow-up.

Exclusion Criteria:

1. Patients who have had other malignant tumors within the past 5 years (excluding cured in situ carcinomas and basal cell skin carcinomas);
2. Patients who have previously received irinotecan treatment;
3. Known allergies to the study drug or its related components;
4. Tumor tissue confirmed by immunohistochemistry to be dMMR status, or confirmed by next-generation sequencing (NGS)/polymerase chain reaction (PCR) to be MSI-H status;
5. Confirmed by next-generation sequencing (NGS)/polymerase chain reaction (PCR) to have BRAF V600E mutation;
6. Participated in other drug clinical trials within four weeks prior to enrollment;
7. Presence of significant gastrointestinal abnormalities during the screening period that, in the investigator's judgment, may affect drug intake, transport, or absorption (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, post-small bowel resection, or total gastrectomy); or history of gastrointestinal perforation and/or fistula; history of peptic ulcer disease within six months prior to the first dose; Intestinal obstruction within 3 months prior to the first dose;
8. History of bleeding, with any severe bleeding event reaching CTCAE 5.0 Grade 3 or higher within 4 weeks prior to screening;
9. Patients with known central nervous system (CNS) metastases or a history of CNS metastases prior to screening. For patients clinically suspected of having CNS metastases, enhanced CT or enhanced MRI must be performed within 28 days prior to randomization to rule out CNS metastases;
10. Patients with hypertension that is not well controlled with single antihypertensive therapy (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); patients with a history of unstable angina; patients newly diagnosed with angina within 3 months prior to screening or who experienced a myocardial infarction event within 6 months prior to screening; Arrhythmia (including QTcF: ≥450 ms in males, ≥470 ms in females) requiring long-term use of antiarrhythmic drugs and New York Heart Association (NYHA) class ≥II heart failure;
11. Urinalysis showing urine protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g;
12. Long-term non-healing wounds or incomplete healing of fractures;
13. Imaging studies showing tumor invasion of important blood vessels or, in the investigator's judgment, a high likelihood of tumor invasion of important blood vessels during treatment, leading to life-threatening hemorrhage;
14. Coagulation abnormalities with a tendency to bleed (must meet the following criteria 14 days prior to enrollment: INR within the normal range without the use of anticoagulants); Patients receiving anticoagulant therapy or vitamin K antagonists such as warfarin, heparin, or their analogues; under the condition that the INR is ≤ 1.5, low-dose warfarin (1 mg orally once daily) or low-dose aspirin (daily dose not exceeding 100 mg) may be used for prophylactic purposes;
15. Patients who have experienced arterial or venous thromboembolic events within the past year, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis (excluding cases where venous thrombosis caused by venous catheterization during prior chemotherapy has been deemed resolved by the investigator), and pulmonary embolism;
16. For female participants: Patients who have not undergone surgical sterilization or are not postmenopausal and refuse to use a medically approved contraceptive method during the study treatment period and for 6 months after the study treatment period; reproductive-age women with a positive serum or urine pregnancy test within 7 days prior to study enrollment, or who are currently breastfeeding. Male participants: Patients who have not undergone surgical sterilization and refuse to use a medically approved contraceptive method during the study treatment period and for 6 months after the study treatment period;
17. Active autoimmune disease or a history of autoimmune disease that may recur;
18. Other patients deemed ineligible for inclusion by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety:The incidence of adverse events | start of treatment until 3-year follow-up
  Proportion of patients experiencing ≥3 grade adverse events (AE) (%);Proportion of patients experiencing AE leading to drug discontinuation (%);Proportion of patients experiencing diarrhea (all grades) (%);Proportion of patients experiencing neutropenia (all grades) (%)

SECONDARY OUTCOMES:
Objective response rate（ORR） | start of treatment until 1-year follow-up
Disease control rate(DCR) | start of treatment until 1-year follow-up
Progression-free survival(PFS) | start of treatment until 2-year follow-up
Overall survival (OS) | start of treatment until 3-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No